CLINICAL TRIAL: NCT04832087
Title: Pediatric Teduglutide Registry: Clinical Use of Teduglutide in Children With Intestinal Failure, a Multicenter Post-marketing Evaluation
Brief Title: Pediatric Teduglutide Registry
Acronym: PTR
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Lissette Jimenez, Co-Director Congenital Enteropathy Program; Attending Physician, Division of Gastroenterology, Hepatology and Nutrition, Boston Children's Hospital
Other Study IDs: P00033923
Record Dates: First submitted 2021-03-29; First posted 2021-04-05 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — teduglutide; ALX-0600

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort A: Participants with SBS who started Teduglutide after FDA approval (May 2019)
  Interventions: Drug: Teduglutide
- Cohort B: Subjects who participated in any of the teduglutide pediatric clinical trial studies (TED-C13-003, TED-C14-006, SHP633-303, or SHP633-304) and subsequently started therapy with teduglutide
  Interventions: Drug: Teduglutide

INTERVENTIONS:
Drug: Teduglutide — Standard of care Teduglutide dosing
  Other Names: Gattex

SUMMARY:
Pediatric specific post-marketing registry to evaluate the long-term safety and efficacy of teduglutide.

DETAILED DESCRIPTION:
This will be a multi-center post-marketing pediatric registry study evaluating the efficacy and safety of teduglutide. This is an observational longitudinal registry of pediatric SBS patients who are using FDA approved teduglutide as per standard of care.

ELIGIBILITY:
Cohort A:

Inclusion Criteria:

1. Diagnosis of SBS defined as intestinal resection for congenital or acquired intestinal disease leading to dependence on PS for 90 days
2. Received teduglutide after FDA approval
3. Age ≥ 1 years and ≤ 18 years at start of teduglutide initiation
4. Weight ≥ 10 kg at start of teduglutide initiation
5. Dependent on PS at the time of teduglutide initiation
6. Subject data for primary outcome (PS energy intake in cal/kg/day) is available for medical chart abstraction at baseline (pretreatment) visit.
7. The subject or guardian signs and dates a written informed consent form and any required privacy authorization and minor provides any assent required prior to enrolment into the registry.

Exclusion Criteria:

1. Participation in the pediatric clinical trial studies of teduglutide (TED-C13-003, TED-C14-006 or SHP633-303, SHP633-304).
2. In the opinion of the investigator, the subject or guardian is at high risk for non-compliance.

Cohort B:

Inclusion Criteria:

1. Diagnosis of SBS defined as intestinal resection for congenital or acquired intestinal disease leading to dependence on PS for 90 days
2. Participated in clinical trial study (TED-C13-003, TED-C14-006) and/or extension study (SHP633-303, SHP633-304)
3. Currently receiving teduglutide
4. The subject or guardian signs and dates a written informed consent form and any required privacy authorization and minor provides any assent required prior to enrolment into the registry.

Exclusion Criteria:

1. In the opinion of the investigator, the subject or guardian is at high risk for non-compliance.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children with SBS on Teduglutide
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Percent change in calories from parenteral support (PS) (Kcal/kg/day) | Up to 3 years
  Maximum percent change in calories (energy intake in kcal/kg/day) from parenteral support relative to pre- treatment (baseline) assessment up to 6 months, 1 year, 2 years and 3 years from start of therapy among Cohort A.

SECONDARY OUTCOMES:
Percent change of (PS) volume (liters/week) | Up to 3 years
  Percent change of PS volume (liters/week) relative to pre-treatment (baseline) assessment up to 6 months, 1 year, 2 years and 3 years from start of therapy among Cohort A
Percent change of PS infusions (number of days/week ) | Up to 3 years
  Percent change of PS infusions (number of days/week relative to pre-treatment (baseline) assessment up to 6 months, 1 year, 2 years and 3 years from start of therapy among Cohort A
Proportion of subjects completely weaned from PS | Up to 3 years
  Number (proportion) of children who wean completely from PS within 6 months, 1 year, 2 years and 3 years from start of therapy among Cohort A.
Adverse Events | Up to 3 years
  Number (proportion) of subjects with adverse events among Cohort A. Number (proportion) of subjects with adverse events among Cohort B.
Weight-for-age Z-score (WAZ) | Up to 3 years
  Mean change in Weight-for-age Z-score (WAZ), relative to pre-treatment (baseline) assessment up to 6 months, 1 year, 2 years and 3 years from start of therapy among Cohort A.
Height-for-age-Z-score (HAZ) | Up to 3 years
  Mean change in Height-for-age-Z-score (HAZ), relative to pre-treatment (baseline) assessment up to 6 months, 1 year, 2 years and 3 years from start of therapy among Cohort A.
Body-Mass-Index Z-score (BMIZ) | Up to 3 years
  Mean change in Body-Mass-Index Z-score (BMIZ), relative to pre-treatment (baseline) assessment up to 6 months, 1 year, 2 years and 3 years from start of therapy among Cohort A.

CONTACTS AND LOCATIONS:
Overall Officials: Lissette Jimenez, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kocoshis SA, Merritt RJ, Hill S, Protheroe S, Carter BA, Horslen S, Hu S, Kaufman SS, Mercer DF, Pakarinen MP, Venick RS, Wales PW, Grimm AA. Safety and Efficacy of Teduglutide in Pediatric Patients With Intestinal Failure due to Short Bowel Syndrome: A 24-Week, Phase III Study. JPEN J Parenter Enteral Nutr. 2020 May;44(4):621-631. doi: 10.1002/jpen.1690. Epub 2019 Sep 8. PMID 31495952
- [Result] Carter BA, Cohran VC, Cole CR, Corkins MR, Dimmitt RA, Duggan C, Hill S, Horslen S, Lim JD, Mercer DF, Merritt RJ, Nichol PF, Sigurdsson L, Teitelbaum DH, Thompson J, Vanderpool C, Vaughan JF, Li B, Youssef NN, Venick RS, Kocoshis SA. Outcomes from a 12-Week, Open-Label, Multicenter Clinical Trial of Teduglutide in Pediatric Short Bowel Syndrome. J Pediatr. 2017 Feb;181:102-111.e5. doi: 10.1016/j.jpeds.2016.10.027. Epub 2016 Nov 15. PMID 27855998